CLINICAL TRIAL: NCT00133614
Title: Prone Positioning in Pediatric Acute Lung Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5336; 5R01NR005336-04 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2005-10-31 (Estimated); Status verified 2005-08

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury | interventions — Prone Position

INTERVENTIONS:
Procedure: Prone Positioning

SUMMARY:
The purpose of this trial is to test the hypothesis that at the end of 28 days, infants and children with acute lung injury treated with prone positioning would have more ventilator-free days than those treated with supine positioning.

DETAILED DESCRIPTION:
Multicenter, randomized, controlled clinical trial conducted from August 28, 2001 to April 23, 2004, of 102 pediatric patients from 7 US pediatric intensive care units aged 2 weeks to 18 years who were treated with supine vs. prone positioning. Randomization was concealed and group assignment was not blinded.

Patients were randomized to either supine or prone positioning within 48 hours of meeting acute lung injury criteria, with those patients in the prone group being positioned within 4 hours of randomization and remaining prone for 20 hours each day during the acute phase of their illness for a maximum of 7 days, after which they were positioned supine. Both groups were treated using lung protective ventilator and sedation protocols, extubation readiness testing, and hemodynamic, nutrition, and skin care guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age >42 weeks post-conceptual age and <18 years of age
* On mechanical ventilation (defined as presence of an endotracheal/tracheostomy tube and currently using ventilator support)
* All of the following in the same 48 hour period:

  * acute pulmonary parenchymal disease (i.e., chest radiograph report of diffuse bilateral pulmonary alveolar infiltrates)
  * mechanical ventilation for at least 1 hour and anticipated need to continue mechanical ventilation for at least 24 hours
  * at least one PaO2/FiO2 ratio <300 (adjusted for barometric pressure: if altitude > 1000m, then PaO2/FiO2 <= 300x(B.P./760), regardless of mean airway pressure)
  * functional arterial catheter for blood gas analysis

Exclusion Criteria:

* Persistent hypotension (defined as systolic blood pressure of 70mmHg+(2x age in years)); i.e. patients requiring either intravenous fluids and/or increases of additional cardiotonic medications every 2 hours
* Active bleeding that requires ongoing blood/fluid volume replacement
* Currently on extracorporeal membrane oxygenation (ECMO)
* Severe chronic lung disease (cystic fibrosis or bronchopulmonary dysplasia)
* Respiratory failure presumed to be the result of cardiac disease
* History of symptomatic or uncorrected congenital heart disease or a right to left intracardiac shunt
* Bone marrow or lung transplant
* Current known diagnosis of any of the following:

  * upper airway disease (i.e., tracheitis, tracheomalacia)
  * reactive airway disease (receiving beta agonists or acute doses of systemic corticosteroids)
  * refractory cerebral hypertension (intracranial pressure [ICP] >20mmHg for 1 hr)
  * neuromuscular respiratory failure (chronic assisted ventilation)
  * spinal instability (uncleared cervical spine)
  * unstable long bone fractures
* Nonpulmonary condition that may be exacerbated by the prone position (for example, osteogenesis imperfecta, craniofacial surgery in the past week)
* Draining abdominal surgical wound
* Pregnancy
* Subject's family/medical team have decided not to provide full support (patient treatment considered futile)
* Enrollment in any other clinical trial within the last 30 days

Ages: 2 Weeks to 18 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 102
Dates: Start 2001-08; Study Completion 2004-04

PRIMARY OUTCOMES:
Prone positioning versus supine positioning in determining ventilator-free days in infants and children

CONTACTS AND LOCATIONS:
Overall Officials: Martha Curley, RN,PhD,FAAN, Principal Investigator — Boston Children's Hospital
Locations (1):
- Childrens Hospital, Boston, Boston, Massachusetts, United States

REFERENCES:
- [Result] Curley MA, Hibberd PL, Fineman LD, Wypij D, Shih MC, Thompson JE, Grant MJ, Barr FE, Cvijanovich NZ, Sorce L, Luckett PM, Matthay MA, Arnold JH. Effect of prone positioning on clinical outcomes in children with acute lung injury: a randomized controlled trial. JAMA. 2005 Jul 13;294(2):229-37. doi: 10.1001/jama.294.2.229. PMID 16014597